CLINICAL TRIAL: NCT03668353
Title: Recombinant SeV-hFGF2 / dF Injection (BF30) Single-dose Therapy in Patients With Peripheral Arterial Occlusive Disease, a Dose Escalation, Safety, Tolerability Phase I Clinical Trial
Brief Title: Recombinant SeV-hFGF2/dF Injection for PAOD
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Salubris Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BF30A101
Record Dates: First submitted 2018-09-08; First posted 2018-09-12 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-09

CONDITIONS: PAOD - Peripheral Arterial Occlusive Disease; PAD; Critical Limb Ischemia
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Intervention Model Description: dose escalation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- treatment 1 (Experimental): Recombinant SeV-hFGF2/dF Injection 2×10 8CIU
  Interventions: Biological: Recombinant SeV-hFGF2/dF Injection
- treatment 2 (Experimental): Recombinant SeV-hFGF2/dF Injection 1×10 9CIU
  Interventions: Biological: Recombinant SeV-hFGF2/dF Injection
- treatment 3 (Experimental): Recombinant SeV-hFGF2/dF Injection 5×10 9CIU
  Interventions: Biological: Recombinant SeV-hFGF2/dF Injection
- treatment 4 (Experimental): Recombinant SeV-hFGF2/dF Injection 1×10 10CIU
  Interventions: Biological: Recombinant SeV-hFGF2/dF Injection

INTERVENTIONS:
Biological: Recombinant SeV-hFGF2/dF Injection — intramuscular injection of investigator drugs
  Other Names: BF30

SUMMARY:
Lower extremity arteriosclerosis obliterans is due to the formation of atherosclerotic plaque in the lower extremities, resulting in the stenosis and occlusion of the artery, leading to chronic ischemia of the limbs. Although bypass surgery and angioplasty ( or interventional therapy ) are effective methods for vascular treatment in patients with PAD to revascularize, a significant proportion of patients with the arterial disease are not eligible for direct arterial surgery. Meanwhile, there are many patients who suffer from diffuse arterial disease or severe peripheral disease not suitable for interventional therapy. Stimulation of arteriogenesis( blood bypassing the occluded arteries through a large number of collateral vessels ) and angiogenesis ( generating new small blood vessels ) have become the focus of research.

Our recombinant SeV-hFGF2/dF injection (R&D code BF30 ) uses the human basic fibroblast growth factor ( FGF2 ) gene to express the target protein FGF2 locally by intramuscular injection. The preparation can efficiently express FGF2 in infected cells and secrete it to the periphery and be fixed in the intercellular substance. Since FGF2 is in the upstream regulatory pathway of VEGF, HGF and other factors, it can regulate the coordinated expression of these cytokines related to the growth and function of new blood vessels, and finally, produce mature blood vessels.

To evaluate the safety ( tolerance), pharmacokinetics (PK), biological activity, and immunogenicity of BF30 in patients with lower extremity arterial occlusive disease, and to explore clinical benefits.

MAIN OBJECTIVE: To evaluate the safety ( tolerability ) of single-dose BF30 in patients with lower extremity arterial occlusive disease, and to provide evidence for the dose of subsequent clinical trials.

Secondary objective: To explore the pharmacokinetics (PK), biological activity, the immunogenicity of BF30, and to initially explore clinical benefits.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-80 years old, weighing > 50kg, with an expected survival of more than 1 year;
* diagnosed as Lower extremity arterial occlusive disease (ASO , DAO , TAO) , and Rutherford grade 2 to 5 (moderate intermittent claudication - mild tissue defect), if both of the subject's limbs have lower extremity arterial ischemic disease, the limb that could not be revascularized or more severe one to study by the investigator;
* Patients are not eligible for revascularization (eg, interventional endovascular treatment or surgery); or patients who have failed previous revascularization treatment;
* For patients who are taking cilostazol, prostaglandins or sarpogrelate for the treatment of lower limb ischemia, a stable dose should be used for at least 1 month before the test drug is injected ;
* Before enrollment, confirmed by DSA or CTA as the superficial femoral artery ( ie, the femoral artery below the branch of the deep femoral artery), one or more stenosis of the radial artery and its lower artery ≥ 75% or occlusion;
* The intended to treat lower extremity ABI ≤ 0.9 ;
* Volunteer to participate in the trial and sign the informed consent form.

Exclusion Criteria:

* Patients with malignant tumors or clinically significant history of a hematological disease, or clinically significant results of tumor screening tests;
* Patients with a history of alcohol or drug abuse in the last 12 months;
* The affected limb may need an amputation in 4 weeks;
* Acute lower extremity arterial ischemic disease or acute progressive disease of lower extremity arterial ischemic disease;
* The index limb has serious infections ( such as cellulitis, osteomyelitis, etc.), distal fascia or bone exposure;
* Cardiac function is classified as grade III or IV heart failure according to the New York Heart Association (NYHA) ;
* Patients with cerebral infarction, cerebral hemorrhage, myocardial infarction, and unstable angina in the past 3 months;
* Type I diabetes patients;
* Poorly controlled hypertension up to three antihypertensive drugs combined, defined as those at screening or baseline testing: systolic blood pressure > 160 mmHg or diastolic blood pressure > 110 mmHg ;
* Patients with grade 3 and above proliferative retinopathy history;
* Currently receiving immunosuppressive agents or radiotherapy and chemotherapy;
* Antiviral drugs, drugs for inhibiting u-PA activity, such as diuretics, amiloride, and suramin, were used within 2 weeks before administration ;
* Subjects included: HIV, hepatitis B, hepatitis C, routine hematology laboratory tests found that patients with significant clinical significance ( hepatitis B virus carriers can be selected); or blood routine, blood biochemistry, liver function, etc. Any of the following abnormalities (if the investigator judges that the abnormality may be caused by the inspection operation, still exists after one retest):

  * TBIL exceeds 1.5 times the normal upper limit or ALT/AST exceeds 2.5 times the upper limit of normal
  * Serum creatinine or urea nitrogen > 1.2 times the upper limit of normal
  * Hemoglobin (Hb) < 8.5 g/dL
  * White blood cell count < 3 × 10 9 /L
  * Platelet count < 75 × 10 9 / L
  * Fasting blood glucose > 13.9 mmol/L
  * HbA1c > 10%
* Donate blood in last 1 month or participate in other intervention clinical trials;
* Childbearing age (male/female) do not agree to adopt recognized effective contraceptives during study treatment and at least 6 months after completion of the study , and / or women of childbearing age who are unwilling or unable to undergo pregnancy tests; pregnancy, Lactating women ( where pregnancy is defined as a positive blood test ) ;
* Other clinically uncontrollable diseases, including but not limited to: a severe liver disease with decompensated cirrhosis, jaundice, ascites or hemorrhagic varices;
* Patients undergoing dialysis;
* a history of allergic to lidocaine, or patients whose may be allergic to the study drug or its components determined by the investigator;
* Other factors that may affect drug safety, effectiveness, and drug metabolism evaluation determined by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-09-05 (Actual); Primary Completion 2020-03-05 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment- Emergent Adverse Events [Safety and Tolerability] | 6 months
  AE incidence, inject site reactions

SECONDARY OUTCOMES:
Maximum Plasma Concentration [Cmax] | 6 months after drug administration
  serum concentration of total RNA
Area Under the Curve [AUC] | 6 months after drug administration
  serum concentration of total RNA
antibody of the SeV | 6 months after drug administration
  Immunogenecity
walking distance | 6 months after drug administration
  walking function
pain scale | 6 months after drug administration
  using VAS scale
Ruthorford staging | 6 months after drug administration
  improvements after study drug use.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No